CLINICAL TRIAL: NCT04518800
Title: Prospective, Open, Single-arm Clinical Study Evaluating the Efficacy and Safety of PEG-rhG-CSF in Secondary Prevention of Nab-Paclitaxel Combined With S-1 in the First-line Treatment of Advanced Pancreatic Cancer
Brief Title: PEG-rhG-CSF in Secondary Prevention of Nab-Paclitaxel Combined With S-1 in Advanced Pancreatic Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Dai, Guanghai, Professor and chief physician, Chinese PLA General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CSPC-JYL-PC-01
Record Dates: First submitted 2020-08-17; First posted 2020-08-19 (Actual); Last update posted 2020-08-19 (Actual); Status verified 2020-08

CONDITIONS: PEG-rhG-CSF; Pancreatic Cancer
Keywords: PEG-rhG-CSF; Secondary Prevention; Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Jin Youli(PEG-rhG-CSF) (Experimental): PEG-rhG-CSF Secondary Prevention：patients with pancreatic cancer who met the eligibility criteria were given secondary prophylactic administration of the Jin Youli(PEG-rhG-CSF).
  Interventions: Drug: Jin Youli(PEG-rhG-CSF)

INTERVENTIONS:
Drug: Jin Youli(PEG-rhG-CSF) — Jin Youli(PEG-rhG-CSF) was given 24 hours after the completion of intravenous infusion of albumin paclitaxel during the treatment period, 6 mg was given to patients with body weight ≥45 kg, and 3 mg was given for body weight <45 kg. Inject once every chemotherapy cycle

SUMMARY:
A prospective, open, single-arm clinical study to evaluate the efficacy and safety of jinyouli（PEG-rhG-CSF） in the first-line treatment of advanced pancreatic cancer with nab-paclitaxel combined with S-1.Chemotherapy regimen: (1) chemotherapy: nab-paclitaxel, 260mg/m2, intravenous infusion for 30 minutes, D1, Q3W. S-1, 80-120mg, PO BID, D1-14, Q3W. (2) patients who met the eligibility criteria were given jinyouli injections 24 hours after the end of intravenous infusion of nab-paclitaxel during the treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years, ≤70 years;
* Patients with Advanced Pancreatic Cancer diagnosed by histopathology，the expected survival time is more than 3 months;
* Neutropenia of ≥2 degree occurred with the nab-paclitaxel + S-1 regimen in the previous cycle.
* KPS score≥70;
* The peripheral blood routine of the patients was normal: ANC ≥ 2.0x10^9/L, platelet count ≥ 90x10^9/L, HB ≥ 80g/L before enrollment, and there was no bleeding tendency;
* Patients volunteered to participate in the trial, signed a written informed consent, willing to be followed up.

Exclusion Criteria:

* There are uncontrollable infections at the moment or systemic antibiotic treatment within 72 h of chemotherapy；
* Any abnormal bone marrow hyperplasia and other abnormal hematopoietic function；
* Patients who had received bone marrow or hematopoietic stem cell transplantation within 3 months；
* Patients with other malignancies that have not been cured or with brain metastases；
* Total bilirubin(TBIL), alanine aminotransferase (ALT) and aspartate aminotransferase (AST) >2.5 ULN, or >5 ULN if there is liver metastasis;
* Serum creatinine (Cr) exceeded the upper limit of normal value；
* Allergic to this product or other biological products derived from genetically engineered escherichia coli；
* Suffering from a mental or nervous system disorder, without self-awareness or coordination；
* Patients expected to have a short survival or have difficulty tolerating chemotherapy；
* Pregnant or lactating female patients；
* Patients using other drugs of the same category or in clinical trials of other drugs；
* Not suitable for participation at investigators' discretion.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-08-18 (Estimated); Primary Completion 2021-08-18 (Estimated); Study Completion 2022-02-18 (Estimated)

PRIMARY OUTCOMES:
Incidence of degree 3-4 neutropenia in each cycle of chemotherapy | last 4 cycles(each cycle is 21 days)
  Incidence of degree 3-4 neutropenia in each cycle of chemotherapy

SECONDARY OUTCOMES:
The incidence of febrile neutropenia in each cycle of chemotherapy | last 4 cycles(each cycle is 21 days)
  Febrile neutropenia (FN) is defined as oral temperature >38.3℃ or continuous measurement of oral temperature >38.1℃ in 1h, with ANC <0.5×10^9/L or expected to be <0.5×10^9/L
Incidence of chemotherapy dose adjustment due to neutropenia in each cycle of chemotherapy | last 4 cycles(each cycle is 21 days)
  Incidence of chemotherapy dose adjustment due to neutropenia in each cycle of chemotherapy
The proportion of patients hospitalized due to neutropenia | last 4 cycles(each cycle is 21 days)
  The proportion of patients hospitalized due to neutropenia
The proportion of patients receiving antibiotics during the entire chemotherapy period. | last 4 cycles(each cycle is 21 days)
  The proportion of patients receiving antibiotics during the entire chemotherapy period.

CONTACTS AND LOCATIONS:
Overall Officials: Guanghai Dai, PhD., Principal Investigator — Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China